CLINICAL TRIAL: NCT03398200
Title: HBO Effects on Blood Count Recovery and Post-transplant Outcomes Following High-dose Therapy and Autologous HSPC Transplantation for Multiple Myeloma
Brief Title: Effects of Hyperbaric Oxygen (HBO) on Blood Count Recovery After Autologous Hematopoietic Stem Cell (HSPC) Transplant for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omar Aljitawi (Other)
Responsible Party: Sponsor-Investigator, Omar Aljitawi, Associate Professor of Hematology/Oncology, University of Rochester
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 70180; UBMT17083 (Other: Wilmot Cancer Institute Clinical Trials Office)
Record Dates: First submitted 2018-01-05; First posted 2018-01-12 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hyperbaric Oxygen Therapy (Experimental): Subjects on the experimental arm will receive 90 minutes of hyperbaric oxygen therapy approximately six hours prior to hematopoietic stem cell infusion.
  Interventions: Biological: Hyperbaric Oxygen Therapy
- No Hyperbaric Oxygen Therapy (Active Comparator): Subjects on the reference arm will not receive hyperbaric oxygen therapy prior to hematopoietic stem cell infusion.
  Interventions: Other: No Hyperbaric Oxygen Therapy

INTERVENTIONS:
Biological: Hyperbaric Oxygen Therapy — The intervention consists of exposure to hyperbaric oxygen at 2.5 atmospheres absolute (ATA) for a total of 2 hours, in a single see-through hyperbaric chamber, breathing 100% oxygen for 90 minutes while subjects are resting in supine position. During the 2 hours, there will be compression and decompression phases for 15 minutes each in which subjects will be breathing compressed environmental air (21% oxygen).
  Arms: Hyperbaric Oxygen Therapy
Other: No Hyperbaric Oxygen Therapy — The reference arm will not receive hyperbaric oxygen therapy prior to hematopoietic stem cell transplant.
  Arms: No Hyperbaric Oxygen Therapy

SUMMARY:
Patients with Multiple Myeloma who are considered for high-dose therapy and autologous transplantation at the bone marrow transplant clinic at the Wilmot Cancer Institute (WCI) will be be approached to participate in this trial. Eligible patients who choose to participate will be randomized so that half receive one hyperbaric oxygen therapy session prior to hematopoetic stem cell infusion and half will not. All subjects will have their blood counts monitored closely and time to count recovery will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent.
* Multiple myeloma diagnosis applying the latest criteria by International Working Group. Patients should have received myeloma-directed induction therapy with appropriate response (partial response or better) in newly diagnosed myeloma patients. Multiple myeloma patients who relapse following induction therapy or following prior autologous hematopoietic stem cell transplant are also eligible as far as remission following their first autologous hematopoietic stem cell transplant lasted 12 months or more.
* Patients who are considered for high-dose therapy and autologous transplantation at the bone marrow transplant clinic at Wilmot Cancer Institute will be screened for eligibility to enroll in this study and if eligible will be approached to participate. Eligible patients will have the chance to tour the hyperbaric oxygen facility prior to signing the consent form.
* Subjects must be ≥ 18 years old and ≤ 75 years old.
* Karnofsky performance status (KPS) of ≥ 70%.
* Adequate hepatic, cardiac and pulmonary function to be eligible for transplant. Minimum criteria include:
* - Alanine aminotransferase (ALT), aspartate aminotransferase (AST): < 4x institutional upper limit of normal (IULN)
* - Total bilirubin: ≤ 2.0 mg/dL
* - Ejection fraction (EF) measured by two-dimensional echocardiography (2D-ECHO) or multigated acquisition (MUGA) scan of ≥ 45%
* - Forced expiratory volume at one second (FEV1), forced vital capacity (FVC), and diffusing capacity of lung for carbon monoxide (DLCO) ≥ 50% of predicted value (corrected to serum hemoglobin)
* - Electrocardiogram (EKG) with no clinically significant arrhythmia.
* Patients should have New York Heart Association (NYHA) Functional Classification, class I or II (No or mild limitation during ordinary activity).
* Patients should be evaluated for fitness for hyperbaric oxygen therapy by a hyperbaric oxygen trained medical professional who is not part of the study team prior to starting preparative regimen.
* Women of child-bearing potential should have a negative urine pregnancy test within 4 weeks of starting preparative regimen.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of therapy. Should a woman or partner become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician and the investigator immediately.
* A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* - Has not undergone a hysterectomy or bilateral oophorectomy; or
* - Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

Exclusion Criteria:

* Pregnant or breastfeeding
* Severe chronic obstructive pulmonary disease requiring oxygen supplementation
* History of spontaneous pneumothorax
* Active ear/sinus infection
* History of sinus or ear surgery, excluding myringotomy or ear tubes
* Claustrophobia
* History of seizures
* Evidence of pneumothorax or significant pulmonary fibrosis on chest imaging
* Prior chest surgery or irradiation
* Patients who had intrathecal chemotherapy within 2 weeks of starting preparative regimen or cranial irradiation within 4 weeks of starting preparative regimen
* Active infection (viral, fungal, and/or bacterial)
* Positive screening for Hepatitis A, B, or C indicating an ongoing infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — Wilmot Cancer Institute
Locations (3):
- United States (3):
  - The University of Kansas Cancer Center, Fairway, Kansas
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Wilmot Cancer Institute, University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
Started | 52 | 47
Completed | 52 | 46
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy | Total
Number analyzed (Participants) | 52 | 47 | 99
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [54 to 67] | 63 [58 to 69] | 62 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 37
  Male | 31 | 31 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 47 | 46 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 46 | 44 | 90
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 52 | 47 | 99

OUTCOME MEASURES:

1. Primary Outcome: Time From Transplant to Neutrophil Count Recovery
Description: Time from transplant to neutrophil recovery was measured as the first day of absolute neutrophil count >=0.5 thou/ul after nadir.
Time Frame: 100 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 52 | 46
days | 12 [12 to 13] | 12 [12 to 13]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Therapy vs No Hyperbaric Oxygen Therapy; Test type: Superiority; p = 0.89, Regression, Cox; 1- degree of freedom (1-df) likelihood ratio test (LRT) in a cell dose stratified Cox model

2. Secondary Outcome: Time From Transplant to Absolute Lymphocyte Recovery
Time Frame: 100 days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 52 | 47
Days | 12 [12 to 13] | 13 [12 to 14]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Therapy vs No Hyperbaric Oxygen Therapy; Test type: Superiority; p = 0.03, Regression, Cox; 1- degree of freedom (1-df) likelihood ratio test (LRT) in a cell dose stratified Cox model

3. Secondary Outcome: Number of Days of Granulocyte Colony-stimulating Factor
Time Frame: 100 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 52 | 47
Days | 6 [5 to 7] | 6 [6 to 6]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Therapy vs No Hyperbaric Oxygen Therapy; Test type: Superiority; p = 0.35, Regression, Cox; 1- degree of freedom (1-df) likelihood ratio test (LRT) in a cell dose stratified Cox model

4. Secondary Outcome: Number of Units of Packed Red Blood Cells Received
Time Frame: 100 days
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 52 | 47
units | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Therapy vs No Hyperbaric Oxygen Therapy; Test type: Superiority; p = 0.77, Regression, Cox; 1- degree of freedom (1-df) likelihood ratio test (LRT) in a cell dose stratified Cox model

5. Secondary Outcome: Length of Hospital Stay
Time Frame: 100 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 44 | 42
Days | 13 [13 to 14] | 14 [13 to 14]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Therapy vs No Hyperbaric Oxygen Therapy; Test type: Superiority; p = 0.50, Regression, Cox; 1- degree of freedom (1-df) likelihood ratio test (LRT) in a cell dose stratified Cox model

6. Secondary Outcome: Percentage of Participants With Progressive Free Survival
Description: A progressive response is defined as follows:
  Increase of > 25% from lowest response value in any one or more of the following:
  Serum M-component and/or (the absolute increase must be > 0.5 g/dL)6 Urine M-component and/or (the absolute increase must be > 200 mg/24 h) Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL Bone marrow plasma cell percentage; the absolute percentage must be > 10%7 Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas Development of hypercalcaemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder
  Anyone who did not have a progressive response was considered as progression free survival.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
Number analyzed (Participants) | 52 | 47
percentage of participants | 91.3 [78.2 to 96.7] | 92.6 [78.6 to 97.6]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Therapy vs No Hyperbaric Oxygen Therapy; Test type: Superiority; p = 0.76, Regression, Cox; 1- degree of freedom (1-df) likelihood ratio test (LRT) in a cell dose stratified Cox model

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | Hyperbaric Oxygen Therapy | No Hyperbaric Oxygen Therapy
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/47
Serious Adverse Events (participants affected / at risk) | 12/52 | 9/47
Other Adverse Events (participants affected / at risk) | 49/52 | 39/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperbaric Oxygen Therapy (N=52) | No Hyperbaric Oxygen Therapy (N=47)
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Sepsis (Infections and infestations) | 4 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Constipation (Immune system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Immune System Disorders - Other, Engraftment Syndrome (Immune system disorders) | 3 | 1
Infections & Infestations - Other, Bacteremia (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 1
Nausea (Immune system disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infections & Infestations - Other, MRSA (Infections and infestations) | 0 | 2
Upper Respiratory Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hyperbaric Oxygen Therapy (N=52) | No Hyperbaric Oxygen Therapy (N=47)
Abdominal Pain (Gastrointestinal disorders) | 18 | 8
Acute Kidney Injury (Renal and urinary disorders) | 1 | 5
ALT Increased (Investigations) | 6 | 9
Anemia (Blood and lymphatic system disorders) | 31 | 23
Anorexia (Metabolism and nutrition disorders) | 14 | 14
Anxiety (Psychiatric disorders) | 4 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
AST Increased (Investigations) | 5 | 6
atrial fibrillation (Cardiac disorders) | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 8
Blood Bilirubin Increased (Investigations) | 5 | 5
Blurred Vision (Eye disorders) | 1 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 7 | 7
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Chills (General disorders) | 7 | 4
Colitis (Gastrointestinal disorders) | 3 | 5
Constipation (Gastrointestinal disorders) | 19 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Creatinine Increased (Investigations) | 3 | 5
Diarrhea (Gastrointestinal disorders) | 37 | 36
Dizziness (Nervous system disorders) | 9 | 12
Dry Mouth (Gastrointestinal disorders) | 2 | 10
Dyspepsia (Gastrointestinal disorders) | 8 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Ear & Labyrinth Disorders - Other, Ear Popping (Ear and labyrinth disorders) | 5 | 0
Ear and Labyrinth Disorders - Other, Ear Pressure (Ear and labyrinth disorders) | 3 | 0
Ear Pain (Ear and labyrinth disorders) | 6 | 0
Edema Limbs (Gastrointestinal disorders) | 12 | 11
Fall (Injury, poisoning and procedural complications) | 3 | 2
Fatigue (General disorders) | 36 | 30
Febrile Neutropenia (Blood and lymphatic system disorders) | 30 | 23
Fever (General disorders) | 3 | 7
Gastrointestinal Disorders - Other, abdominal crampin (Gastrointestinal disorders) | 4 | 3
Headache (Nervous system disorders) | 13 | 12
Hematuria (Renal and urinary disorders) | 3 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 5 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 4
Hypertension (Vascular disorders) | 14 | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 22 | 18
Hypocalcemia (Metabolism and nutrition disorders) | 40 | 37
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 20 | 27
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 14
Hyponatremia (Metabolism and nutrition disorders) | 1 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 30 | 33
Hypotension (Vascular disorders) | 13 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Immune System Disorders - Other, Engraftment Syndrome (Immune system disorders) | 4 | 1
Infections & Infestations - Other, Bacteremia (Infections and infestations) | 4 | 5
Insomnia (Psychiatric disorders) | 17 | 15
Leukopenia (Blood and lymphatic system disorders) | 40 | 37
Lung Infection (Infections and infestations) | 3 | 0
Lymphopenia (Blood and lymphatic system disorders) | 36 | 34
Metabolism & nutritional disorders - other, insufficient oral intake (Metabolism and nutrition disorders) | 1 | 3
Mucositis Oral (Gastrointestinal disorders) | 22 | 17
Myalgia (General disorders) | 5 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 42 | 36
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 42 | 38
Non-Cardiac Chest Pain (General disorders) | 1 | 5
Pain (General disorders) | 1 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 7
Peripheral Sensory Neuropathy (Nervous system disorders) | 10 | 11
Pruitus (Skin and subcutaneous tissue disorders) | 0 | 3
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 | 2
Renal & Urinary Disorders - Other, Dysuria (Renal and urinary disorders) | 3 | 2
Respiratory, Thoracic & Mediastinal Disorders - Other, runny nose (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 3
Sinus Tachycardia (Cardiac disorders) | 16 | 11
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 41 | 39
Thromboembolic Event (Vascular disorders) | 5 | 1
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 22 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT03398200/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT03398200/ICF_001.pdf